CLINICAL TRIAL: NCT06311669
Title: Comparative Study Between Isolated Iliac Vein Stenting Versus Concomitant Iliac Vein Stenting With Pelvic Vein Embolization in Patients With Pelvic Venous Insufficiency Secondary to Nonthrombotic Iliac Vein Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29409010104798
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-12

CONDITIONS: Nonthrombotic Iliac Vein Lesions; Pelvic Congestive Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isolated iliac vein stenting (Active Comparator)
  Interventions: Procedure: iliac vein stenting
- Concomitant iliac vein stenting with pelvic vein embolization (Active Comparator)
  Interventions: Procedure: iliac vein stenting; Procedure: pelvic vein embolization

INTERVENTIONS:
Procedure: iliac vein stenting — patients will undergo left common iliac vein stenting according to diameter measurements using balloon-mounted stents.
Procedure: pelvic vein embolization — embolization of pelvic veins by injection of left ovarian vein or parauterine veins pelvic escape points using sandwich technique of detachable or pushable coils and polidocanol 3 %.
  Arms: Concomitant iliac vein stenting with pelvic vein embolization

SUMMARY:
The aim of the study is to compare between Isolated Iliac vein stenting vs Concomitant Iliac vein stenting with pelvic vein embolization in patients with Pelvic Venous Insufficiency secondary to Nonthrombotic iliac vein lesions

DETAILED DESCRIPTION:
* Type of Study: Prospective randomized 2 arms clinical trial
* Study Setting: Ain Shams University hospitals
* Study Period: 6 months
* Sample Size: 20 patients
* Study Population Female patients walking in or referred to the out-patient clinic at Ain Shams University Specialized Hospitals or El-Demerdash University Hospitals with symptoms of pelvic venous insufficiency.
* Inclusion Criteria:

  1. Female Patients
  2. Child-baring period (18-50)
  3. Patients with type 2 Pelvic congestion (defined as venous substitute pathology secondary to stenosis or obstruction in a draining vein according to Greiner classification of pelvic congestion) (Milka Greiner., et al 2017)
  4. Patients with Nonthrombotic iliac vein lesions confirmed by Duplex with Peak Systolic Velocity (PSV) ratio between stenotic and pre stenotic segment > 2.5.
  5. CEAP Classification C 0,1,2

Exclusion Criteria:

1. Pregnancy
2. Breast-feeding
3. Menopause
4. Patients with type 1 Pelvic congestion (defined as reflux pathology secondary to valvular or parietal venous anomaly without pelvic or supra-pelvic obstruction to venous flow according to Greiner classification of pelvic congestion) (Milka Greiner., et al 2017)
5. Patients with type 3 Pelvic congestion (defined as local extrinsic cause responsible for pelvic venous anomaly according to Greiner classification of pelvic congestion) (Milka Greiner., et al 2017)
6. CEAP Classification C 3,4,5

   * Sampling Method Convenient sample
   * Ethical Considerations An informed consent will be taken from every patient prior to having the procedure to document having their approval for both, having the procedure and participating in the study with emphasis that their medical treatment will not be affected by their refusal of participation according to approved standards to ethical committee of Ain Shams University.
   * Study Tools 20 patients will be randomly divided into 2 equal groups (A and B) Written informed consent. Full history taking with pelvic pain assessment (by onset, course, duration, site, character, radiation, aggravating and reliving factors, severity, timing, associated symptoms) and other pelvic symptoms, urinary symptoms or piles assessment guided by The Pelvic Venous Clinical Severity Score (PVCSS) giving the patient a score.

Clinical Assessment and examination of the patients including tenderness in left iliac fossa and vulvar varicosities, after exclusion of gynaecological causes confirmed by Gynaecology.

Full Lab investigations (complete blood count, coagulation profile, serum creatinine).

Radiological investigations:

1. Combined pelviabdominal and transvaginal ultrasound to determine the diameter and the reflux of the ovarian veins, internal iliac veins and para uterine veins with diameter of ovarian vein > 6mm and para uterine vein > 5mm, also the criteria to diagnose Nonthrombotic iliac vein lesions with Peak Systolic Velocity (PSV) ratio between stenotic and pre stenotic segment > 2.5.
2. CT Venography. All patients will undergo Multiplaner venogram via ultrasound guided puncture through popliteal vein, Great Saphenous Vein (GSV), Common femoral vein to view the left common iliac vein and to view the pelvic escape points after cannulation of the left renal vein Group A patients will undergo left common iliac vein stenting according to diameter measurements using balloon-mounted stents.

Group B patients will undergo concomitant iliac vein stenting and embolization of pelvic veins by injection of left ovarian vein or parauterine veins pelvic escape points using sandwich technique of detachable or pushable coils and polidocanol 3 %.

Analysis of the results. Statistical Analysis: Collected data will be tabulated and analyzed using SPSS (IBM SPSS Statistics for Mac, Version 25.0. IBM Corp., Armonk, NY). Chi-square test and ANOVA will be used for categorical data, t-test will be used to compare mean values of non-categorical data between both groups, suitable graphs and figures will be plotted to demonstrate relevant statistics.

Primary end point:

Clinical improvement of pain and pelvic symptoms according to the Pelvic Venous Clinical Severity Score (PVCSS)

ELIGIBILITY:
Inclusion Criteria:

- 1) Female Patients 2) Child-baring period (18-50) 3) Patients with type 2 Pelvic congestion (defined as venous substitute pathology secondary to stenosis or obstruction in a draining vein according to Greiner classification of pelvic congestion) (Milka Greiner., et al 2017) 4) Patients with Nonthrombotic iliac vein lesions confirmed by Duplex with Peak Systolic Velocity (PSV) ratio between stenotic and pre stenotic segment > 2.5.

5) CEAP Classification C 0,1,2

Exclusion Criteria:

* 1) Pregnancy 2) Breast-feeding 3) Menopause 4) Patients with type 1 Pelvic congestion (defined as reflux pathology secondary to valvular or parietal venous anomaly without pelvic or supra-pelvic obstruction to venous flow according to Greiner classification of pelvic congestion) (Milka Greiner., et al 2017) 5) Patients with type 3 Pelvic congestion (defined as local extrinsic cause responsible for pelvic venous anomaly according to Greiner classification of pelvic congestion) (Milka Greiner., et al 2017) 6) CEAP Classification C 3,4,5

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement of pain and pelvic symptoms according to the Pelvic Venous Clinical Severity Score (PVCSS) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman Salem, Study Director — Professor of vascular surgery, faculty of medicine Ainshams university
Locations (1):
- Ainshams University, Cairo, Egypt